CLINICAL TRIAL: NCT05849727
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Trial to Evaluate the Efficacy and Safety of TQH3821 Tablets in Patients With Treated Rheumatoid Arthritis
Brief Title: A Clinical Study of TQH3821 Tablets in the Treatment of Treated Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per sponsor request.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH3821-II-01
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQH3821 tablets 200 mg (Experimental): Oral administration of TQH3821 tablets 200 mg, twice a day for 24 weeks.
  Interventions: Drug: TQH3821 tablets 200 mg
- TQH3821 tablets matching placebo (Placebo Comparator): The placebo group was taken orally until the end of week 12. At the end of week 12, the placebo group was switched to the oral administration of TQH3821 tablets 200 mg until the end of week 24.
  Interventions: Drug: TQH3821 tablets 200 mg; Drug: TQH3821 tablets matching placebo

INTERVENTIONS:
Drug: TQH3821 tablets 200 mg — TQH3821 is a Interleukin-1 Receptor-Associated Kinase 4 (IRAK4) inhibitor.
Drug: TQH3821 tablets matching placebo — TQH3821 tablets matching placebo without active substance.
  Arms: TQH3821 tablets matching placebo

SUMMARY:
To evaluate the efficacy and safety of TQH3821 in treated patients with moderate-to-severe active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent;
* Male and female, ≥18 years old and ≤70 years old (subject to the date of signing the informed consent);
* The diagnosis meets the rheumatoid arthritis (RA) classification criteria jointly established by the American College of Rheumatology (ACR) and the European Alliance against Rheumatism (EULAR) in 2010, for at least 3 months ;
* Moderate to severe active RA was defined by the following criteria: joint swelling ≥6 (based on 66 joints), joint tenderness ≥6 (based on 68 joints), Disease activity score 28-C-reactive protein (DAS28-CRP) ≥3.2, and CRP>10mg/L or erythrocyte sedimentation rate (ESR) >28mm/h;
* At least 12 weeks of treatment with methotrexate (dose 7.5 to 25 mg/ week) and stable dose (7.5 to 25 mg/ week) ≥4 weeks prior to initial administration of the study drug (oral stable dose methotrexate will be continued as background therapy during the trial);
* The subjects can attend the study visit on time and complete the visit;

Exclusion Criteria:

* 8 weeks before baseline examination, subjects underwent joint surgery or received intraarticular glucocorticoid therapy at the joint sites evaluated in this study;
* Patients with rheumatoid arthritis with joint functional activity grade Ⅳ or confined to a wheelchair or bed;
* Current or previous inflammatory joint diseases other than RA and other autoimmune venereal diseases;
* Patients with lung diseases deemed unsuitable for the study by the investigator;
* Cardiovascular and cerebrovascular abnormalities;
* Abnormal thyroid function;
* Subjects with a history or suspected demyelinating disease of the central nervous system;
* Have any type of active malignant tumor or have a history of malignant tumor;
* Presence of active Mycobacterium tuberculosis (TB) infection or latent TB infection without appropriate treatment;
* Have any acute or chronic active infectious disease;
* There are serious poorly controlled diseases;
* People with active hepatitis, or hepatitis B surface antigen (HBsAg) positive, hepatitis B core antibody (HBcAb) positive + hepatitis B virus (HBV) DNA positive, or hepatitis C virus (HCV) antibody-positive;
* History of human immunodeficiency virus (HIV) infection, or positive HIV serological results at screening, and positive antibodies to treponema pallidum during screening;
* Subjects who had suffered a severe trauma, fracture, or surgical procedure within 8 weeks prior to screening, or who were expected to require major surgical procedures during the study period;
* Female subjects who are pregnant or lactating;
* Those who received live attenuated vaccine within 28 days before the start of treatment, inactivated vaccine within 7 days, or planned vaccination during the study period;
* The subject has any medical condition that may affect oral drug absorption, gastrectomy or gastrointestinal disease of clinical significance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 20 (ACR20) improvement | Evaluated at week 12.
  Proportion of patients with ACR20 at week 12.

SECONDARY OUTCOMES:
American College of Rheumatology 20 (ACR20) improvement | Evaluated at week 4, 8, 18, and 24.
  Proportion of patients with ACR20.
American College of Rheumatology 50 (ACR50) improvement | Evaluated at week 4, 8, 12, 18, and 24.
  Proportion of patients with ACR20.
C-reactive protein (CRP) | Evaluated at week 4, 8, 12, 18, and 24.
  Changes in C-reactive protein (CRP) relative to baseline.
Erythrocyte sedimentation rate (ESR) | Evaluated at week 4, 8, 12, 18, and 24.
  Changes in erythrocyte sedimentation rate (ESR) relative to baseline.
66 joint swelling counts (SJC) | Evaluated at week 4, 8, 12, 18, and 24.
  Change in the number of 66 joint swelling relative to baseline.
68 joint tenderness counts (TJC) | Evaluated at week 4, 8, 12, 18, and 24.
  Change in the number of 68 joint tenderness numbers (TJC) relative to baseline.
Disease activity score 28-C-reactive protein (DAS28-CRP) | Evaluated at week 4, 8, 12, 18, and 24.
  Changes in disease activity score DAS28 -CRP relative to baseline.
Patient's visual analogue score (PVAS) | Evaluated at week 4, 8, 12, 18, and 24.
  PVAS is a questionnaire to evaluate joint pain in subjects with scores from 0 to 10, where 0 means no pain and 10 means the worst pain.
Patient's global assessment (PtGA) | Evaluated at week 4, 8, 12, 18, and 24.
  PtGA is a questionnaire to evaluate arthritis score by patient's overall assessment, with scores from 0 to 10, where 0 means very good and 10 means very poor.
Physician's global assessment (PhGA) | Evaluated at week 4, 8, 12, 18, and 24.
  PhGA is a questionnaire to evaluate arthritis score by physician's overall assessment, with scores from 0 to 10, where 0 means very good and 10 means very poor.
Health Assessment questionnaire-Disability Index (HAQ-DI) | Evaluated at week 4, 8, 12, 18, and 24.
  HAQ-DI is a questionnaire to evaluate quality of life of subjects with scores from 0 to 3, 0 means easy and 3 means very difficult.
Incidence of adverse events | Baseline up to 28 weeks.
  Incidence of adverse events after administration.
Severity of adverse events | Baseline up to 28 weeks.
  Severity of adverse events after administration.

CONTACTS AND LOCATIONS:
Locations (34):
- China (34):
  - Bozhou People's Hospital, Bozhou, Anhui
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - The Peking University People's Hospital, Beijing, Beijing Municipality
  - The Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Qiqihar, Qiqihar, Heilongjiang
  - Anyang District Hospital of Puyang City, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Xiangya Third Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - China-japan Friendship Hospital of Jilin University, Changchun, Jilin
  - Central Hospital of Jinzhou, Jinzhou, Liaoning
  - Heze Municipal Hospital, Heze, Shandong
  - Yantaishan Hospital of Yantai, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Tongji Hospital, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of PLA Air Force Medical University, Xi’an, Shanxi
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Wenling First People's Hospital, Taizhou, Zhejiang
  - Taizhou Central Hospital Taizhou University Hospitai, Taizhou, Zhejiang
  - Yuyao People's Hospital, Yuyao, Zhejiang